CLINICAL TRIAL: NCT01719289
Title: Cluster Randomised Controlled Trial of a Primary-care Based Intervention to Improve Depressive Symptoms of Pregnant Women in Sao Paulo, Brazil
Brief Title: Efficacy of a Program for the Management of Depression in Pregnant Women in Primary Care in São Paulo, Brazil
Acronym: PROGRAVIDA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Sao Paulo General Hospital (Other)
Collaborators: Conselho Nacional de Desenvolvimento Científico e Tecnológico (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CNPq 575320/2008-7
Record Dates: First submitted 2012-10-29; First posted 2012-11-01 (Estimated); Last update posted 2012-11-01 (Estimated); Status verified 2012-10

CONDITIONS: Depression
Keywords: depression; problem solving
MeSH Terms: conditions — Depression

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- PROGRAVIDA (Experimental): All women in this arm receive a stepped-care program for depression based on psycho-education and problem solving techniques.
  Interventions: Behavioral: PROGRAVIDA
- Treatment as usual (No Intervention): Primary health care professionals in charge of prenatal care are notified by the research team about all women with depression receiving pre-natal care and included in the trial. Primary health care professionals decide how to treat these women without any interference from the research team.

INTERVENTIONS:
Behavioral: PROGRAVIDA — Women in the intervention group receive a program based on psycho-education and problem solving techniques, delivered by a nurse assistant at the women's homes. The program comprises 8 sessions, 6 during pregnancy and 2 after delivery. Intensity of depressive symptoms is assessed using the PHQ-9, at the beginning of the sessions. Women with severe depression are referred to the family doctor and are assessed for the need of antidepressant medication.
  Arms: PROGRAVIDA

SUMMARY:
Background: depression during pregnancy is an important problem for public health. It has direct consequences for the affected woman, her children and family, and is a strong predictor of post-partum depression. In developing countries depression during pregnancy is highly common, and usually unrecognized and untreated.

Aim: to evaluate the effectiveness and cost-effectiveness of an intervention delivered by nurse assistants in the management of pregnant women with depression in primary care clinics that adopt the Family Health Strategy in Sao Paulo, Brazil.

Method: PROGRAVIDA is a cluster randomized controlled trial with pregnant women with depression attending pre-natal care in 12 Primary Care Units with Family Health Program, covering an area of 400,000 inhabitants in Sao Paulo, Brazil. The intervention follows a stepped-care approach and is delivered by health professionals working at the primary care unit responsible by the care of the women. All women from the intervention group receive a program based on psycho-education and problem solving techniques, delivered by a nurse assistant at the women's homes. The program comprises 8 sessions, 6 during pregnancy and 2 after delivery. Intensity of depressive symptoms is assessed using the PHQ-9, at the beginning of the sessions. Women with severe depression are referred to the family doctor and are assessed for the need of antidepressant medication. The control group receives routine care. The primary outcome is remission of depressive symptoms 4-months after the inclusion in the study. Secondary outcomes include remission of depressive symptoms at 6 months after delivery. Women are also assessed for socioeconomic and household characteristics, social support and obstetric complications. The effectiveness and cost-effectiveness of the intervention will be assessed with intention-to-treat analysis, using the clinical outcome and the assessment of quality of life (EQ-5D) four months after inclusion in the trial.

DETAILED DESCRIPTION:
Despite the high prevalence of depressive disorders in pregnancy and puerperium and the possible negative consequences of these frames for women, children and family, there are still very scarce evidence on the effectiveness of interventions of low cost and viable, that can be made available on the net of Primary Health Care in Brazil and other middle or low income countries.

The main objective of this study is to evaluate the effectiveness of a depression management program, simple and low cost, delivered by nurse assistants, in reducing symptoms of depression in pregnant women treated in primary care clinics that adopt the Family Health Strategy (FHS) in São Paulo, compared to routine care. We will also assess the cost-effectiveness of this intervention.

We are conducting a community cluster randomized trial with pregnant women with symptoms of depression, attending antenatal care in primary care clinics that adopt the FHS in São Paulo. Participating clinics (12) were randomly allocated to have their nurse assistants receiving training and supervision to perform a program for management of depression among pregnant women (experimental group) or to offer routine care (control group).

ELIGIBILITY:
Inclusion Criteria:

Pregnant women attending antenatal care in selected primary care clinics with Family Health Programs, who score a PHQ-9>=5 just after the first antenatal consultation or around the 20th week of pregnancy.

Exclusion Criteria:

Moderate to high suicidal risk (assessed with a standardised protocol),

* Ongoing psychiatric treatment,
* Not able to understand Portuguese.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2011-03; Primary Completion 2013-11 (Estimated); Study Completion 2014-09 (Estimated)

PRIMARY OUTCOMES:
Patient Health Questionnaire (PHQ-9) | 4 months after inclusion in the study
  PHQ-9 score=<4 will be considered success

SECONDARY OUTCOMES:
PHQ-9 | 6 months after delivery
  PHQ-9 score=<4 will be considered success
General Quality of life (EQ-5D) | 4 months after inclusion and 6 months after delivery
  The instrument contains 2 parts: a descriptive part that evaluates five domains (mobility, self care, usual activity, discomfort / pain and anxiety / depression). In this section a person assesses the current health on a scale 1-3 (none, moderate and severe). The respondent also makes self-evaluation through visual scale grading their health from 0 (worst possible) to 100 (best possible).

CONTACTS AND LOCATIONS:
Overall Officials: Paulo R Menezes, PhD, Principal Investigator — University of Sao Paulo; Marcia Scazufca, PhD, Study Director — University of Sao Paulo
Locations (1):
- Faculdade de Medicina da Universidade de Sao Paulo, São Paulo, São Paulo, Brazil